CLINICAL TRIAL: NCT00862095
Title: A Randomized Controlled Trial of Medical Therapies for Chronic Post-Traumatic Headaches
Brief Title: Medical Therapies for Chronic Post-Traumatic Headaches
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate enrollment, insufficient funds to continue enrollment
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay C. Erickson, Chief, Neurology Service, Madigan Army Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 208075
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Propranolol; Amitriptyline; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo
- Propranolol (Experimental): Propranolol (target dose 80 mg a day)
  Interventions: Drug: Propranolol
- Topiramate (Experimental): Topiramate (target dose 100 mg a day)
  Interventions: Drug: Topiramate
- Amitriptyline (Experimental): Amitriptyline (target dose 50 mg a day)
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Placebo — Every month for 3 months
  Arms: Placebo
Drug: Propranolol — target does 80 mg per day for 3 months
  Other Names: Inderal
  Arms: Propranolol
Drug: Amitriptyline — Target does of 50 mg per day for 3 months
  Other Names: Elavil
  Arms: Amitriptyline
Drug: Topiramate — Target dose 100 mg a day for 3 months
  Other Names: Topamax
  Arms: Topiramate

SUMMARY:
To determine if propranolol, amitriptyline, or topiramate decreases headache frequency in patients with chronic post-traumatic headaches.

DETAILED DESCRIPTION:
A total of 240 patients meeting International Classification of Headache Disorders (ICHD) diagnostic criteria for chronic post-traumatic headaches will be enrolled. Subjects will be recruited from the Neurology Clinic at Madigan Army Medical Center. Study participants will be U.S. Army soldiers who sustained a mild traumatic head injury while deployed to a combat theater resulting in chronic post-traumatic headaches. Subjects will be randomized to placebo, propranolol (target dose 80 mg a day), amitriptyline (target dose 50 mg a day), or topiramate (target dose 100 mg a day) for 3 months.

The primary outcome measure will be the mean number of headache days per month on the third month of treatment. Secondary outcome measures will include the proportion of subjects with at least a 25% reduction in headache frequency, headache severity (0-10 scale), headache duration (hours), headache-related disability (measured by the Headache Impact Test and Migraine Disability Assessment Scale), PTSD symptom checklist score, and medication side effects and tolerability.

ELIGIBILITY:
Inclusion criteria:

1. Patient meets ICHD criteria for chronic post-traumatic headaches (see below).
2. Patient is 18-50 years old.
3. Patient has experienced 6 or more days of headache per month for each of the last 2 months.
4. Patient has full capacity to provide informed consent.
5. Patient will be available for all study-related visits over the next 4 months.
6. Patient must be eligible to receive care at Madigan Army Medical Center

International Classification of Headache Disorders (version 2) diagnostic criteria for chronic post-traumatic headaches attributed to mild head injury:

1. Headaches beginning within 1 week of mild traumatic head injury.
2. Headaches persisting > 3 months after head trauma.
3. Head trauma with all of the following:

   * no loss of consciousness or loss of consciousness < 30 minutes
   * Glasgow Coma Score (GCS) 13-15
   * symptoms or signs diagnostic of concussion

Exclusion criteria:

1. Patient has another headache disorder not attributable to head trauma which accounts for at least half of the patient's headache episodes.
2. Patient is currently taking propranolol, amitriptyline, or topiramate for any reason.
3. Patient previously tried propranolol, amitriptyline, or topiramate for headache treatment.
4. Patient started a new treatment for headache prevention within the last 6 weeks. Prophylactic treatments initiated prior to 6 weeks ago are allowed as long as the dose or regimen is stable. Medications for aborting acute headaches are also allowed.
5. Patient previously tried more than two medications for headache prevention.
6. Patient is using narcotic analgesics on average more than 10 days a month.
7. Patient has a medical condition or is taking a medication that is considered a contraindication for propranolol, topiramate, or amitriptyline. Medical conditions include liver disease, renal impairment, cardiac dysrhythmias, untreated thyroid disease, orthostatic hypotension, asthma requiring treatment with inhalers, glaucoma, kidney stones, insulin-requiring diabetes, or pregnancy.
8. Patient has known hepatic, renal, or cardiac disorders.
9. Patient drinks on average more than two servings of alcohol (2 oz hard liquor, 5 oz wine, 12 oz beer) per day or more than 3 servings at one time on a weekly basis.
10. Patient has abnormalities on baseline EKG.
11. Patient has major depression defined as a score >15 on the Patient Health Questionnaire-9.
12. Patient is pregnant, planning to become pregnant in the next year, or is a female of reproductive potential who is not using a reliable form of birth control.
13. Patient has cognitive impairment defined as mini-mental status exam score <27.
14. SBP < 90, HR < 50, or HR > 100.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Headache days per month on the third month of treatment | Monthly for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Erickson, MD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States